CLINICAL TRIAL: NCT01782807
Title: Ovarian Function After Hysterectomy With or Without Fimbriectomy or Salpingectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Lion Poles, Deputy Director of Kaplan Medical Center, Kaplan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: kmc0029-11
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2011-06

CONDITIONS: Ovarian Function Insufficiency
Keywords: Ovarian function; Hysterectomy; Salpingectomy; Anti mullerian hormone
MeSH Terms: interventions — Salpingectomy; Sterilization, Tubal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hysterectomy (No Intervention): Hysterectomy without oophorectomy or salpingectomy
- Hysterctomy with salpingectomy or fimbriectomy (Experimental): Salpingectomy or Fimbriectomy
  Interventions: Procedure: Salpingectomy or Fimbriectomy

INTERVENTIONS:
Procedure: Salpingectomy or Fimbriectomy
  Arms: Hysterctomy with salpingectomy or fimbriectomy

SUMMARY:
The impact of Hysterectomy with preservation of the ovaries on ovarian function has long been controversial. studies have shown conflicting data regarding ovarian function after simple Hysterectomy.

In recent years, there is a growing evidence that Salpingectomy or Fimbriectomy may have preventive value reducing Ovarian and Primary Peritoneal carcinoma, but the safety and the consequences regarding ovarian function have yet to be established.

The aim of this study is to evaluate ovarian function after Hysterectomy alone Vs. Hysterectomy combined with salpingectomy or fimbriectomy

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing Hysterectomy for Benign In dication (eg. Uterus Myomatous) before menopause

Exclusion Criteria:

* Menopause
* known or suspected malignancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Ovarian function | 60 days post-operative
  ovarian function measured by FSH , AMH and follicule count on ultra-sound

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

REFERENCES:
- [Background] Maseela T, Scheele R. [Hysterosalpingectomy. A contribution to the prevention of primary tubal neoplasms]. Fortschr Med. 1980 Jun 5;98(21):818-22. German. PMID 7409710
- [Background] Zalel Y, Lurie S, Beyth Y, Goldberger S, Tepper R. Is it necessary to perform a prophylactic oophorectomy during hysterectomy? Eur J Obstet Gynecol Reprod Biol. 1997 May;73(1):67-70. doi: 10.1016/s0301-2115(97)02702-4. PMID 9175692
- [Background] Morse AN, Hammer RA, Walter AJ, Baker S, Magtibay PM. Does hysterectomy without adnexectomy in patients with prior tubal interruption increase the risk of subsequent hydrosalpinx? Am J Obstet Gynecol. 2002 Dec;187(6):1483-5; discussion 1485-6. doi: 10.1067/mob.2002.130212. PMID 12501050
- [Background] Farquhar CM, Sadler L, Harvey SA, Stewart AW. The association of hysterectomy and menopause: a prospective cohort study. BJOG. 2005 Jul;112(7):956-62. doi: 10.1111/j.1471-0528.2005.00696.x. PMID 15957999
- [Background] Riedel HH, Lehmann-Willenbrock E, Semm K. Ovarian failure phenomena after hysterectomy. J Reprod Med. 1986 Jul;31(7):597-600. PMID 3746790
- [Background] Bulent Tiras M, Noyan V, Ozdemir H, Guner H, Yildiz A, Yildirim M. The changes in ovarian hormone levels and ovarian artery blood flow rate after laparoscopic tubal sterilization. Eur J Obstet Gynecol Reprod Biol. 2001 Dec 1;99(2):219-21. doi: 10.1016/s0301-2115(01)00410-9. PMID 11788175